CLINICAL TRIAL: NCT00927732
Title: BRD 06/2-D (Quidam) "Evaluation of the Interest of Oral Hydroquinidine Administration to Treat Patients With Brugada Syndrome, High Cardiac Arrhythmic Risk and Implanted With an Implantable Cardioverter Defibrillator"
Brief Title: Hydroquinidine Versus Placebo in Patients With Brugada Syndrome
Acronym: Quidam
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment, a lot of premature study discontinuations
Sponsor: Nantes University Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06/2-D
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Brugada Syndrome
Keywords: Brugada; hydroquinidine; ventricular arrhythmia; patients with Brugada syndrome, high cardiac arrhythmic risk and implanted with an implantable cardioverter defibrillator
MeSH Terms: conditions — Brugada Syndrome | interventions — hydroquinidine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydroquinidine (Experimental): As it is a cross-over study, patient will taken treatment 1 for 18 months (ex: hydroquinidine) and then treatment 2 (placebo in this case) for 18 months.
  Interventions: Drug: hydroquinidine
- capsules of sugar (Placebo Comparator): As it is a cross-over study, patient will taken treatment 1 for 18 months (ex: hydroquinidine) and then treatment 2 (placebo in this case) for 18 months.
  Interventions: Drug: placebo (sugar)

INTERVENTIONS:
Drug: hydroquinidine — capsules of 300 mg LP, 1 or 2 or 3 times per day : frequency will be determined by tests after patient inclusion before her/his randomization
  Other Names: Hydroquinidine is commercialized as Serecor
  Arms: hydroquinidine
Drug: placebo (sugar) — capsules of placebo have same design and color than capsules of hydroquinidine except for their content as they contain sugar and not hydroquinidine
  Arms: capsules of sugar

SUMMARY:
The specific aim of this study is to determine whether hydroquinidine administration can prevent heart from appearance of ventricular arrhythmia detected by the automatic implantable defibrillator (ICD).

DETAILED DESCRIPTION:
During this double-blind randomized cross-over study, patient will receive during 18 months treatment 1 (hydroquinidine or placebo) and, after 7 days of wash-out, patient will receive treatment 2 (meaning for example hydroquinidine if treatment 1 was placebo). Time length before arisen of an appropriate shock registered on the defibrillator (meaning due to ventricular arrhythmia) will be assessed during treatment 1 period and treatment 2 period.We hypothesized that hydroquinidine administration will enhance time length before arisen of an appropriate shock and thus mean that hydroquinidine administration can prevent heart from appearance of ventricular arrhythmia. Patient's defibrillator recordings will be analysed every 6 months plus when patient experiences an ICD shock. If the shock delivered by the ICD is appropriate and happens during treatment 1 period, patient will switch to treatment 2 period after 7 days of wash-out. If the shock delivered by the ICD is appropriate and happens during treatment 2 period, study will be finished for this patient.Before starting the study, each patient will test which dose of hydroquinidine she/he requires to have an hydroquinidine concentration in her/his blood included between 3 and 6 µmol/L.

Planned enrollment: 200 subjects (60 being symptomatic with histories of aborted sudden cardiac death or of ventricular fibrillation, 70 being symptomatic with histories of syncope considered as of arrhythmic origin, 70 being asymptomatic with a spontaneous type 1 ECG and a positive electrophysiological exploration)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult (at least 18 years of age)
* Informed consent form signed
* Subject affiliated to French health insurance (Sécurité Sociale)
* Type 1 Brugada syndrome either symptomatic or asymptomatic
* Not pregnant, taking oral contraceptive measure if able to procreate
* If patient with asymptomatic type 1 Brugada, electrophysiological exploration must be positive at study inclusion
* No current intake of "betablocking" medicine used in cardiac insufficiency (bisoprolol, carvedilol, metoprolol)
* No current myasthenia
* No current treatment with halofantrine, pentamidine, moxifloxacin
* No current treatment with some neuroleptics
* Known hypersensitivity to hydroquinidine
* Intolerance to fructose, syndrome of glucose or galactose malabsorption, deficit in sucrase isomaltase- Cardiac insufficiency
* Histories of "torsades de pointe"
* Intake of medicine giving "torsades de pointe"

Exclusion Criteria:

* Subject not fulfilling inclusion criteria
* Subject being before study entry under hydroquinidine treatment but either at a dose > 3 capsules per day or at a dose of 1, 2 or 3 capsules per day but with a plasmatic hydroquinidine concentration >6µmol/L or <3 µmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To determine whether hydroquinidine enhances time length before arisen of an appropriate shock registered on the automatic implantable defibrillator (meaning due to ventricular arrhythmia) | 3 years after patient randomization

SECONDARY OUTCOMES:
To evaluate number and frequency of inappropriate shock with and without hydroquinidine | 3 years after patient randomization
To evaluate the number of tachycardia or of ventricular fibrillations detected by the defibrillator but not having required any treatment | 3 years after patient randomization
To evaluate number of syncope reported by the patient but for which no ventricular arrhythmias has been detected by the defibrillator | 3 years after patient randomization
To evaluate the number and frequency of adverse events appeared under hydroquinidine treatment | 3 years after patient randomization
To evaluate interest of the electrophysiological exploration for determining chances of success of an hydroquinidine | 3 years after patient randomization

CONTACTS AND LOCATIONS:
Overall Officials: V Probst, Pr, Principal Investigator — CHU NANTES - Hôpital Laennec; JM Dupuis, Dr, Study Chair — University Hospital, Angers; JS Hermida, Pr, Study Chair — CHU AMIENS; M Haissaguerre, Pr, Study Chair — University Hospital, Bordeaux; J Mansourati, Pr, Study Chair — CHU BREST; P Defaye, Dr, Study Chair — University Hospital, Grenoble; S Kacet, Pr, Study Chair — CHRU LILLE; P Chevallier, Pr, Study Chair — Hospices Civils de Lyon; JC Deharo, pr, Study Chair — CHU MARSEILLE; JM Davy, Pr, Study Chair — University Hospital, Montpellier; N Sadoul, Pr, Study Chair — CHU NANCY; A Leenhardt, Pr, Study Chair — CHU PARIS LARIBOISIERE; A Amiel, Dr, Study Chair — CHU Poitiers; P Mabo, Pr, Study Chair — CHU Rennes; M Chauvin, Pr, Study Chair — CHU STRASBOURG; D Babuty, Pr, Study Chair — CHU Tours; P Maury, Dr, Study Chair — University Hospital, Toulouse
Locations (17):
- France (17):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Grenoble, Grenoble
  - CHRU Lille, Lille
  - CHU Lyon, Lyon
  - AP-HM Marseille, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - AP-HP Paris Lariboisière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours